CLINICAL TRIAL: NCT04392167
Title: Advanced Angle-Resolved Low Coherence Interferometry (a/LCI) Systems for Improved Clinical Utility: An a/LCI-Optical Coherence Tomography (OCT) Pilot Study
Brief Title: a/LCI-OCT Pilot in Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00090173_1; R01CA210544 (NIH)
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- a/LCI-OCT Imaging of the Esophagus (Experimental)
  Interventions: Device: a/LCI-OCT imaging probe; Procedure: esophageal biopsy

INTERVENTIONS:
Device: a/LCI-OCT imaging probe — a/LCI and OCT imaging measurements of several locations in the esophagus
Procedure: esophageal biopsy — biopsies of esophageal tissue imaged by a/LCI-OCT probe

SUMMARY:
This study will test a newly developed dual modality probe, including optical coherence tomography (OCT) and angle-resolved low-coherence interferometry (a/LCI), in the human esophagus to determine 1) whether adequate tissue contact can be attained by the probe to acquire high quality images, and 2) to identify if these images can discern whether the imaged tissue is squamous or Barrett's Esophagus (BE) epithelium. This pilot study will test the operating characteristics of the probe and collect data for further optimization of the a/LCI-OCT device.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to University of North Carolina (UNC) for routine care upper endoscopy
* Meet one of the following criteria:

  1. Current dysplastic or non-dysplastic Barrett's Esophagus of any length OR,
  2. History of dysplastic or non-dysplastic Barrett's Esophagus after treatment with endoscopic eradication therapy (EET) OR,
  3. Normal asymptomatic controls without any history of dysplastic Barrett's Esophagus
* Aged 18 to 80
* Able to read, comprehend, and understand the informed consent document

Exclusion Criteria:

* Prior esophageal surgery (uncomplicated nissen fundoplication OK)
* Pregnant women
* Unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wax, Ph.D., Principal Investigator — Professor
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terry NG, Zhu Y, Rinehart MT, Brown WJ, Gebhart SC, Bright S, Carretta E, Ziefle CG, Panjehpour M, Galanko J, Madanick RD, Dellon ES, Trembath D, Bennett A, Goldblum JR, Overholt BF, Woosley JT, Shaheen NJ, Wax A. Detection of dysplasia in Barrett's esophagus with in vivo depth-resolved nuclear morphology measurements. Gastroenterology. 2011 Jan;140(1):42-50. doi: 10.1053/j.gastro.2010.09.008. Epub 2010 Sep 18. PMID 20854820

RESULTS

PARTICIPANT FLOW:
Groups:
- a/LCI-OCT Imaging of the Esophagus: All participants who were able to swallow the a/LCI-OCT probe had a/LCI-OCT imaging of the esophagus. These participants then also had biopsies of the esophageal tissue that was imaged by the a/LCI-OCT probe.
Period: Overall Study
Arm/Group | a/LCI-OCT Imaging of the Esophagus
Started | 37
Completed | 31
Not Completed | 6
Not completed — unable to swallow a/LCI-OCT probe | 6

BASELINE CHARACTERISTICS:
Arm/Group | a/LCI-OCT Imaging of the Esophagus
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant did not report age.
  years
    number analyzed (Participants) | 36
    (all) | 65.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant did not report sex.
  Participants
    number analyzed (Participants) | 36
    Female | 8
    Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37
Stage of Barrett's Esophagus [Count of Participants; unit: Participants]
  non-dysplastic Barrett's Esophagus | 12
  Barrett's Esophagus with low grade dysplasia | 7
  Barrett's Esophagus with high grade dysplasia | 16
  history of Barrett's Esophagus with CEIM (complete eradication of intestinal metaplasia) | 1
  normal asymptomatic control without history of Barrett's Esophagus | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correctly Identified Positive (Dysplastic) Biopsies
Description: Sensitivity of the a/LCI-OCT probe to detect dysplasia as measured by percentage of correctly identified positive biopsies. The a/LCI-OCT measurement of mean nuclear size was compared with a pre-determined threshold of mean nuclear size (11.84 microns from Terry et al study) to categorize biopsy samples as dysplastic or non-dysplastic.
Time Frame: day 1
Measure: Number; unit: percentage of correct identifications
Units Other Than Participants: positive biopsies
Arm/Group | a/LCI-OCT Imaging of the Esophagus
Number analyzed (Participants) | 3
Number analyzed (positive biopsies) | 7
percentage of correct identifications | 100.0

2. Primary Outcome: Percentage of Correctly Identified Negative (Non-Dysplastic) Biopsies
Description: Specificity of the a/LCI-OCT probe to detect absence of dysplasia as measured by percentage of correctly identified negative biopsies. The a/LCI-OCT measurement of mean nuclear size was compared with a pre-determined threshold of mean nuclear size (11.84 microns from Terry et al study) to categorize biopsy samples as dysplastic or non-dysplastic.
Time Frame: day 1
Measure: Number; unit: percentage of correct identifications
Units Other Than Participants: negative biopsies
Groups:
- a/LCI-OCT Imaging of the Esophagus: All participants who were able to swallow the a/LCI-OCT probe had a/LCI-OCT imaging of the esophagus, with measurements in at least 5 locations. These participants then also had biopsies of the esophageal tissue that was imaged by the a/LCI-OCT probe.
Arm/Group | a/LCI-OCT Imaging of the Esophagus
Number analyzed (Participants) | 22
Number analyzed (negative biopsies) | 43
percentage of correct identifications | 93.0

3. Secondary Outcome: Percentage of Participants With Adequate Tissue Contact to Acquire a High Quality Image
Description: percentage of participants that had adequate tissue contact to acquire high quality a/LCI-OCT images
Time Frame: day 1
Measure: Number; unit: percentage of participants
Arm/Group | a/LCI-OCT Imaging of the Esophagus
Number analyzed (Participants) | 37
percentage of participants | 83.8

ADVERSE EVENTS:
Time Frame: 1 week
Description: Participants were contacted 1 week after a/LCI-OCT imaging to assess any adverse events.
Arm/Group | a/LCI-OCT Imaging of the Esophagus
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 22/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | a/LCI-OCT Imaging of the Esophagus (N=37)
sore throat (Surgical and medical procedures) | 20
throat tightness / trouble swallowing (Surgical and medical procedures) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT04392167/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT04392167/ICF_000.pdf